CLINICAL TRIAL: NCT05627206
Title: The Impact of PM+For Moms Intervention on Improving Mother's Mental Health in Zambia (PM+FM)
Acronym: PM+FM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Innovations for Poverty Action (Other)
Responsible Party: Principal Investigator, Irene Falgas Bague, Post-Doctoral Research Collaborator, Swiss Tropical & Public Health Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PM+FMZam
Record Dates: First submitted 2022-11-07; First posted 2022-11-25 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Depressive Symptoms; Anxiety; Trauma, Psychological
Keywords: women; low-resourced settings; psychosocial intervention
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Trauma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Problem Management + For Moms

INTERVENTIONS:
Behavioral: Problem Management + For Moms — Psychosocial intervention conducted by a trained Wellbeing-Community health worker. Adapted from Problem Management +, thinking healthy and Strong Minds-Strong Communities intervention to target women with small children and mental health symptoms living in low-resourced settings. Combines several evidence-based strategies such us psychoeducational, motivational interviewing, cognitive restructuring and relaxation exercises. Organized in 10 weekly sessions (8 individual 2 in group) provided in-person, by phone or virtually.
  Arms: Intervention

SUMMARY:
CMHD are particularly prevalent among women, posing a major threat to their own and their children's wellbeing.

Despite the high prevalence of CMHD and the existence of effective treatments, interventions supporting women living in low-resourced settings remain limited.

This study builds on a parent study (Zamcharts NCT03991182), which identified a high prevalence of women with anxiety and/or depression. We propose to design, test, and validate a community-based intervention nested within the public primary health system in Zambia, to identify and treat women with mild-to-severe CMHDs.

ELIGIBILITY:
Inclusion Criteria:

* Women participating in ZamCharts parent study
* SRQ-20 >7 (clinically significant symptoms of depression or/anxiety),
* not planning to move within the next 6 months,
* with capacity to consent
* not receiving current mental health care.

Exclusion Criteria:

* Women with active suicidal ideation (determined by Paykel=4 OR 5),
* severe substance use (ACOK-SUD >4),
* mania or psychotic symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Mental health symptoms. SRQ-20 | Change between Baseline (at enrollment) and 6 months after enrollment
  20 items measuring risk of common mental health problem.
Feasibility of the study | Assessed 4 months after enrollment
  % of 1 or more sessions completed. Qualitative feedback from participants and providers.
Acceptability | Assessed 4 months after enrollment
  % of participants completing more than 6 sessions. Qualitative feedback from participants and providers.

SECONDARY OUTCOMES:
Change in Mental health symptoms. PSYCHLOPS | Used for the pre-post treatment analysis. Change between Baseline (at enrollment) and 4 months after enrollment
  Psychological Outcome Profiles (5 items)
Functionality | Used for the pre-post treatment analysis. Change between Baseline (at enrollment) and 4 months after enrollment
  WHO-DAS2
World Bank's Toolkit and Inventory | Used for the pre-post treatment analysis. Change between Baseline (at enrollment) and 4 months after enrollment
  Selected measures from the World Bank Toolkit to address mother-child interactions and child early development.
Change in Anxiety and Depression symptoms. | Used for the pre-post treatment analysis. Change between Baseline (at enrollment) and 4 months after enrollment
  HSCL-25. 10 questions anxiety, 15 depression; (α = 0.90).

CONTACTS AND LOCATIONS:
Locations (1):
- Innovatations for Poverty Action, Lusaka, Zambia

REFERENCES:
- [Derived] Fink G, Melero-Dominguez M, Chembe M, de Vernisy-Romero D, Tembo T, Billima T, Paul R, Alegria M, Parkerson D, Rockers PC, Banda Z, Lungu G, Sikazwe D, Falgas-Bague I. Feasibility and acceptability of the Problem Management for Moms programme for improving maternal mental health in Zambia: an open-label trial. Lancet Psychiatry. 2024 Dec;11(12):965-974. doi: 10.1016/S2215-0366(24)00256-6. Epub 2024 Nov 5. PMID 39515361
- [Derived] Falgas-Bague I, Melero-Dominguez M, de Vernisy-Romero D, Tembo T, Chembe M, Lubozha T, Paul R, Parkerson D, Rockers PC, Sikazwe D, Fink G. Testing the feasibility, acceptability, and exploring trends on efficacy of the problem management plus for moms: Protocol of a pilot randomized control trial. PLoS One. 2024 Jan 5;19(1):e0287269. doi: 10.1371/journal.pone.0287269. eCollection 2024. PMID 38181004